CLINICAL TRIAL: NCT05551481
Title: 2 Year Follow-up of Indirect Resin Composite Restorations Luted With Different Adhesive Resin Cement: A Randomized Clinical Trial
Brief Title: Follow-up of Indirect Restorations Luted With Different Adhesive Resin Cement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, yeldaerdem, Dr., Istanbul Medipol University Hospital
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: Indirect Resin Composite
Record Dates: First submitted 2022-08-19; First posted 2022-09-22 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Dental Restoration Failures
Keywords: indirect composite
MeSH Terms: interventions — Variolink

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In Group A,(Variolink II, Ivoclar Vivadent). (Experimental): In Group A, the onlays and overlays were luted adhesively with etch and rinse, dual cure resin cement (Variolink II, Ivoclar Vivadent).
  Interventions: Procedure: To evaluate the clinical performance of indirect resin composite restorations, which were luted with two different resin cement, in posterior teeth for up to 2 years.
- In Group B, (Relyx U200, 3M ESPE). (Active Comparator): In Group B the onlays and overlays were luted using a self-adhesive resin cement (Relyx U200, 3M ESPE).
  Interventions: Procedure: To evaluate the clinical performance of indirect resin composite restorations, which were luted with two different resin cement, in posterior teeth for up to 2 years.

INTERVENTIONS:
Procedure: To evaluate the clinical performance of indirect resin composite restorations, which were luted with two different resin cement, in posterior teeth for up to 2 years. — resin cement (Variolink II, Ivoclar Vivadent)-self-adhesive resin cement (Relyx U200, 3M ESPE)
  Other Names: restorations made of laboratory-processed- luted using an etch and rinse resin cement (Variolink II, Ivoclar Vivadent) and 22 onlay restorations (Group B) were luted using a self-

SUMMARY:
Objective: To evaluate the clinical performance of indirect resin composite restorations, which were luted with two different resin cement, in posterior teeth for up to 2 years.

Methods: From February 2017 to May 2017, a total of 43 patients (21 men, 22 women; mean age.), received 48 onlay restorations made of laboratory-processed indirect composite (Gradia, GC, Japan). 27 onlay restorations (Group A) were luted using an etch and rinse resin cement (Variolink II, Ivoclar Vivadent) and 22 onlay restorations (Group B) were luted using a self-adhesive resin cement (Relyx U200, 3M ESPE). Patients were followed until May 2019. Two independent calibrated examiners evaluated the restorations at 3-time points: 2 weeks after placement (baseline), 6 months, and then annually, using the modified USPHS/FDI criteria.

DETAILED DESCRIPTION:
Study design The ethical committee of Istanbul Medipol University approved this clinical study. Patients were given written informed consent to participate before treatment and agreed to a recall program at baseline 2 weeks, 6 months, and thereafter annually. All restorative procedures were carried out by one experienced dentist from the Department of Restorative Dentistry at Istanbul Medipol University.

Inclusion and exclusion criteria

Patients in need of removal of old large amalgam restorations or having extensive caries lesions were recruited for the study. Inclusion and exclusion criteria were as follows:

Adults of at least 18 years of age, with good oral hygiene, having an antagonist tooth in occlusion, being mentally in a good state to provide written consent to participate in the clinical study, and willing to attend the scheduled follow-up appointments. Exclusion criteria included the presence of teeth with severe periodontal problems, high caries risk, and bruxism.

Cavities were prepared according to common principles, which included an occlusal reduction of 1.5-2 mm with a wide isthmus and rounded occlusal-axial angles, and an axial wall of 1.5 mm in thickness. Where possible, the gingival margins were prepared entirely in enamel at the cemento-enamel junction, and cavities for overlays included both buccal and lingual/palatal cusps. Both cavity types (onlays and overlays) were prepared with rounded internal angles, with a divergence of 6-15° between the walls and margins with a 90° cave surface.

Full-arch impressions were made with a single impression/double mixing technique using polyether material (Impregum Penta H Duoso, 3M ESPE, Minn, USA) cavity preparations were provisionalized for 1 week with photo-polymerized provisional material (Clip, Voco, Cuxhaven, Germany). All onlays were definitively inserted within 1 week after impression. After the removal of provisional restorations, the teeth were thoroughly cleaned with a prophylaxis brush and pumice.

After adjustment when needed, the restorations were luted adhesively under a rubber dam, employing a total-etch system in group A. The prepared teeth were initially cleaned with pumice slurry and etched with 35% phosphoric acid gel (Ultra-etch, Ultradent, South Jordan, UT, USA). The dentin adhesive system (Syntac Classic, Ivoclar Vivadent, Liechtenstein) was then applied uniform and gently air thinned. The internal surface of the restorations was silanized (Monobond S, Ivoclar Vivadent), waited for its reaction for 60 s and the solvent was evaporated with oil-free compressed air. The onlays and overlays were luted adhesively with etch and rinse, dual cure resin cement (Variolink II, Ivoclar Vivadent). In Group B were luted using a self-adhesive resin cement (Relyx U200, 3M ESPE).

Excess resin cement was removed in all cases with an explorer, a brush, and dental floss interproximally. Each only surface was light-cured for 40 s with a polymerization light (Elipar Highlight, 3M Espe, Seefeld, Germany). After placement and removal of the rubber dam, static and dynamic occlusion was adjusted using fine grit diamond burs, then inlays were finished with disks and strips (Sof-Lex, 3M Dental Products, St. Paul, MN, USA).

ELIGIBILITY:
Inclusion criteria Patients in need of removal of old large amalgam restorations or having extensive caries lesions were recruited for the study.

Adults of at least 18 years of age, with good oral hygiene, having an antagonist tooth in occlusion, being mentally in a good state to provide written consent to participate in the clinical study, and willing to attend the scheduled follow-up appointments.

Exclusion criteria Exclusion criteria included the presence of teeth with severe periodontal problems, high caries risk, and bruxism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18-65
Enrollment: 40 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Endocrowns FDI evaluation | 2 year
  this clinical trial aimed to evaluate posterior teeth restored with indirect resin composites and compare clinical performances of two resin cement (one etch and rinse and one self-adhesive) 2 weeks and 6, 12, 24 months, and 5 years after the luting of indirect resin composite restorations using the modified USPHS/FDI criteria.

SECONDARY OUTCOMES:
Aesthetic :Functional :Biological :Vitality-resin cement | 2 weeks and 6, 12 months and 2 year
  Surface luster-Surface staining-Colour stability and translucency-Anatomic form.Fracture and retention-Marginal adaptation-Wear -Proximal contact-Patient's viewFracture and retention-Marginal adaptation-Wear -Proximal contact-Patient's view.Postoperative hypersensitivity-Recurrent of caries, erosion, abfraction-Tooth integrity-Vitality-resin cement

CONTACTS AND LOCATIONS:
Overall Officials: yelda erdem hepsenoglu, Study Chair — Medipol University
Locations (1):
- Yelda Erdem Hepsenoglu, Istanbul, Turkey (Türkiye)